CLINICAL TRIAL: NCT03369054
Title: Determining the Feasibility and Effectiveness of Psychotherapy for Transgender Clients: A Randomized Controlled Trial
Brief Title: Psychotherapy Trial With Transgender Clients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017-0816; A171600 (Other: UW Madison); EDUC\COUNSELING PSYCH (Other: UW Madison)
Record Dates: First submitted 2017-11-27; First posted 2017-12-11 (Actual); Last update posted 2019-12-24 (Actual); Status verified 2019-01

CONDITIONS: Transgender Persons, M01.777.500
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Minority Stress (Experimental): The (MST) condition will include a psychoeducation session on minority stress for all participants during the initial assessment session prior to their first psychotherapy session. Prior to attending each of the 12 psychotherapy sessions during their electronic assessment (filling out the OQ-45 on Qualtrics on a computer provided by the study team), patients will be prompted to report up to three minority stress experiences over the previous week in the survey tool (which the therapists will not see). They will be prompted by their therapist to discuss these experiences within their psychotherapy sessions (for example, "Would you like to discuss any of the minority stress experiences you've had over the week?").
  Interventions: Behavioral: Minority Stress Treatment
- Treatment as Usual (Active Comparator): Treatment-as-usual (TAU) will occur as any usual 12-week treatment. The therapists will be encouraged to discuss any of the presenting concerns reported by patients and supervision will include usual care.
  Interventions: Behavioral: Treatment As usual

INTERVENTIONS:
Behavioral: Minority Stress Treatment — The (MST) condition will include a psychoeducation session on minority stress for all participants during the initial assessment session prior to their first psychotherapy session. Prior to attending each of the 12 psychotherapy sessions during their electronic assessment (filling out the OQ-45 on Qualtrics on a computer provided by the study team), patients will be prompted to report up to three minority stress experiences over the previous week in the survey tool (which the therapists will not see). They will be prompted by their therapist to discuss these experiences within their psychotherapy sessions (for example, "Would you like to discuss any of the minority stress experiences you've had over the week?").
  Arms: Minority Stress
Behavioral: Treatment As usual — Treatment-as-usual (TAU) will occur as any usual 12-week treatment. The therapists will be encouraged to discuss any of the presenting concerns reported by patients and supervision will include usual care.
  Arms: Treatment as Usual

SUMMARY:
Transgender and gender diverse (TGD) individuals are at an increased risk for mental health concerns, including anxiety, trauma-based distress, depression, self-harm, and suicidality. Quantitative and qualitative studies have shown that support appears to mediate mental health concerns, but to date, there have been zero psychotherapy studies focusing on transgender and gender diverse patients. The NIH has noted that TGD patients are considered to be a "health disparities population," indicating that there is considerable research to support prevention and reduction in mental health disparities for this population.

There are two aims to the current study-Aim 1: investigate the feasibility of conducting a psychotherapy randomized controlled trial for transgender and gender diverse populations, and Aim 2: longitudinally investigate the impact of minority stress interventions on well-being for transgender and gender diverse patients.

First, it is hypothesized that this study will demonstrate feasibility regarding recruitment of transgender and gender diverse patients and that patients from both groups will report treatment acceptability. We also hypothesize that patients will report more acceptability for treatments that are focused on minority stress interventions. It is hypothesized that individuals in both the Minority Stress Treatment (MST) group and Treatment as Usual (TAU) group will both show improvements in well-being, but that the MST group will demonstrate larger effects in outcomes.

No known published studies have focused on minority stress psychotherapy interventions for transgender and gender diverse populations. The findings from the proposed study will provide a multitude of information regarding longitudinal psychotherapy interventions focusing on minority stress that will inform future treatment manuals and larger, multi-site studies.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 or older
* Fluent in written and spoken English
* Willingness to participate in pre/post/session-by-session assessments and 12 ----Individual psychotherapy treatment sessions
* Individual identifies as transgender, trans, or non-binary (or somewhere along the gender minority spectrum).

Exclusion Criteria:

* Under 18 years old
* Reports current, unmanaged psychotic symptoms or symptoms requiring immediate inpatient treatment (e.g., hallucinations, delusions, threatening immediate suicidal behaviors)
* Currently engaging in psychotherapy
* Cannot attend therapy on Tuesdays from 2-7pm
* Individuals who lack the capacity to provide consent will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — All participants must identify as transgender or gender non conforming
Enrollment: 20 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-01-10 (Actual); Study Completion 2019-01-10 (Actual)

PRIMARY OUTCOMES:
Measuring Weekly Change in the Outcome Questionnaire 45; Lambert et al., 2013 | Week 1, Week 2, Week 3, Week 4, Week 5, Week 6, Week 7, Week 8, Week 9, Week 10, Week 11, Week 12, 3 months, 9 months (within 6 months of study completion)
  Measures overall mental health (symptom distress, interpersonal relations, social role). This is a 45-item likert scale. The total score ranges from 0 - 180 and includes a cutoff score of 63 or more (indicating symptoms of clinical distress). Higher scores suggest more symptoms of distress and difficulties in relationships. For symptom distress, scores range from 0-100 and the clinical cutoff score is 36 or more. For interpersonal relations, scores range from 0-44 and has a cutoff score of 15 or more. For social role, the range is 0-36 and includes a cutoff score of 12 or more. For all scales, higher scores indicate more distress. All scales are summed.
Measuring 3 month and 9 month Change in the Outcome Questionnaire 45; Lambert et al., 2013 | Prior to Week 1 (within 2 weeks of Week 1), 3 months, 9 months (within 6 months of study completion)
  Measures overall mental health (symptom distress, interpersonal relations, social role). This is a 45-item likert scale. The total score ranges from 0 - 180 and includes a cutoff score of 63 or more (indicating symptoms of clinical distress). Higher scores suggest more symptoms of distress and difficulties in relationships. For symptom distress, scores range from 0-100 and the clinical cutoff score is 36 or more. For interpersonal relations, scores range from 0-44 and has a cutoff score of 15 or more. For social role, the range is 0-36 and includes a cutoff score of 12 or more. For all scales, higher scores indicate more distress. All scales are summed.

SECONDARY OUTCOMES:
Measuring 3 month and 9 month Change in the World Health Organization WHOQOL-BREF Quality of Life Assessment (WHOQOL-BREF); Power, 1998 | Prior to Week 1 (within 2 weeks of Week 1), 3 months after starting Week 1, and 9 months after Week 1
  This scale measures quality of life based on functioning (physical, psychological, social, and environment). The scale includes 26 questions on a likert scale. Scores range from 26-130 and are summed. Higher scores indicate higher quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Budge, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Budge SL, Tebbe EA, Love D. The Development and Pilot Testing of a Minority Stress Psychoeducation Tool for Transgender and Nonbinary People. Transgend Health. 2024 Jun 17;9(3):275-279. doi: 10.1089/trgh.2022.0038. eCollection 2024 Jun. PMID 39109257
- [Derived] Budge SL, Guo E, Mauk E, Tebbe EA. The development of an observational coding scheme to assess transgender and nonbinary clients' reported minority stress experiences. Psychotherapy (Chic). 2021 Jun;58(2):288-300. doi: 10.1037/pst0000368. PMID 34410793
- [Derived] Budge SL, Sinnard MT, Hoyt WT. Longitudinal effects of psychotherapy with transgender and nonbinary clients: A randomized controlled pilot trial. Psychotherapy (Chic). 2021 Mar;58(1):1-11. doi: 10.1037/pst0000310. Epub 2020 Jun 22. PMID 32567869